CLINICAL TRIAL: NCT00821977
Title: Efficacy and Long-Term Safety of Vildagliptin as Monotherapy in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLAF237B2201
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; Vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Vildagliptin Dose 1 (Experimental)
  Interventions: Drug: Vildagliptin
- Vildagliptin Dose 2 (Experimental)
  Interventions: Drug: Vildagliptin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin
  Arms: Vildagliptin Dose 1
Drug: Vildagliptin
  Arms: Vildagliptin Dose 2
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a 2-3 period parallel group study with an adaptive element in Type 2 diabetes patients receiving vildagliptin as monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age at Visit 1
* Drug naïve patients with T2DM diagnosed at least 2 months prior to Visit 1
* HbA1c ≥ 7.0 % and ≤ 10.0% at Visit 1
* Body Mass Index (BMI) in the range of 22-45 kg/m2 at Visit 1

Exclusion Criteria:

* Pregnant or lactating female
* FPG ≥ 270 mg/dL (≥15 mmol/L)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Measure: To evaluate the efficacy of vildagliptin as monotherapy in patients with T2DM by assessing changes in HbA1c from baseline to 24 weeks. | 24 weeks

SECONDARY OUTCOMES:
Measure: To evaluate the efficacy of vildagliptin as monotherapy in patients with T2DM as measured by changes in fasting plasma glucose from baseline to 24 weeks | 24 weeks
Measure: To evaluate the safety and tolerability of vildagliptin compared to placebo over 24 weeks of treatment as monotherapy in patients with T2DM | 24 weeks
Measure: To evaluate the long-term safety and tolerability of vildagliptin over the entire study duration as monotherapy in patients with T2DM | 76 weeks
Measure: To evaluate the body weight change from baseline with vildagliptin compared to placebo after 24 weeks of treatment as monotherapy in patients with T2DM | 24 weeks

CONTACTS AND LOCATIONS:
Locations (176):
- United States (141):
  - Advanced Clinical Research, Pell City, Alabama
  - Horizon Clinical Research Associates, PLLC, Gilbert, Arizona
  - Vista Medical Research, Inc, Mesa, Arizona
  - Clinical Research Advantage, Mesa, Arizona
  - Hope Clinical Research, Phoenix, Arizona
  - Anasazi Internal Medicine, Phoenix, Arizona
  - Tatum Ridge Internal Medicine, Phoenix, Arizona
  - Paradigm Clinical, Tucson, Arizona
  - Tucson Clinical Research, Tucson, Arizona
  - Medical Investigations, Inc., Little Rock, Arkansas
  - Paul W. Davis, MD, Pine Bluff, Arkansas
  - Sall Research Medical Center, Artesia, California
  - Associated Pharmaceutical Research, Buena Park, California
  - Providence Research, Burbank, California
  - Burbank - Lovelace Scientific Resources, Inc., Burbank, California
  - Lucita M. Cruz, M.D., Inc., Norwalk, California
  - California Research Foundation, San Diego, California
  - Ritchken and First MDs, San Diego, California
  - San Diego Sports Medicine Research and Family Care, San Diego, California
  - Crest Clinical Trials, Santa Ana, California
  - NuLife Clinical Research, Inc., Santa Ana, California
  - Westside Arthritis and Metabolism Center, Santa Monica, California
  - Center for Clinical Trials of San Gabriel, West Covina, California
  - Colorado Springs Health Partners, Pc, Colorado Springs, Colorado
  - Express Care Clinical Research, Colorado Springs, Colorado
  - Cherry Creek Family Practice, Denver, Colorado
  - Metro Clinical Research, Littleton, Colorado
  - Complete Family Care, Northglenn, Colorado
  - Clinical Therapeutics Corp, Coral Gables, Florida
  - Fort Lauderdale, Florida
  - South Florida Clinical Research Center, Miramar, Florida
  - Pines Research, LLC, Pembroke Pines, Florida
  - Well Pharma Medical Research, South Miami, Florida
  - Southern Clinical Research, Augusta, Georgia
  - Rockdale Medical Research, Conyers, Georgia
  - North Georgia Medical Research Institute, Ellijay, Georgia
  - Perimeter North Medical Research, Roswell, Georgia
  - JMG CIinical Research, Alton, Illinois
  - Fox Valley Clinical Research, Aurora, Illinois
  - American Health Network, Indianapolis, Indiana
  - Mercy Family Medicine, Mason City, Iowa
  - Associates Research, Inc, Lansing, Kansas
  - Health Science Research Center, Pratt, Kansas
  - Cotton O'neil Clinic, Topeka, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Dolby Research, LLC, Baton Rouge, Louisiana
  - Bruce Samuels LLC, Covington, Louisiana
  - Gulf Coast Research, LLC, Lafayette, Louisiana
  - Crescent City Clinical Research Center, Metairie, Louisiana
  - The Family Doctors, Shreveport, Louisiana
  - Maine Centers for Endocrinology & Diabetes, Scarborough, Maine
  - Michigan Hypertension Center, Chelsea, Michigan
  - Genesys Integrated Group Practice, PC, Flint, Michigan
  - Borgess Heart Institute-Borgess Research Institute, Kalamazoo, Michigan
  - NISUS Research Northern MI Hospital, Petoskey, Michigan
  - Spence Medical Research Center, LLC, Pinckney, Michigan
  - Southwestern Medical Clinic, PC, Stevensville, Michigan
  - Belzoni Clinical Research, Belzoni, Mississippi
  - Gulfside Clinical Research, Gulfport, Mississippi
  - Mississippi Medical Research, LLC, Picayune, Mississippi
  - Woodlake Research, Chesterfield, Missouri
  - Midwest Pharmaceutical Research Inc., City of Saint Peters, Missouri
  - Midwest Pharmaceutical Research, Inc., City of Saint Peters, Missouri
  - Truman Medical Center & Univ Physician Associates, Kansas City, Missouri
  - Ozark Mountains Medical Research, Ozark, Missouri
  - Ozark Medical-Surgical Associates, Ltd., Springfield, Missouri
  - ClinVest Research, Springfield, Missouri
  - Patient's First Health Care, Washington, Missouri
  - Physician Research Collaboration, Lincoln, Nebraska
  - Fallbrook Family Health Center, Lincoln, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Heartland Clinical Research, Inc., Omaha, Nebraska
  - Desert Endocrinology Clinical Research Center, Henderson, Nevada
  - Clinical Research Center of NV, Las Vegas, Nevada
  - Palm Medical Research Center, Las Vegas, Nevada
  - Joslin Diabetes Center, Nashua, New Hampshire
  - Shore Health Group, Toms River, New Jersey
  - Physicians Research Center, Toms River, New Jersey
  - The Endocrine Group, LLP, Albany, New York
  - Endwell Family Physician, Endwell, New York
  - North Shore Diabetes and Endocrine Associates, New Hyde Park, New York
  - Mezitis Education & Research Institute, New York, New York
  - Cornerstone Medical Center, Burlington, North Carolina
  - Kernodle Clinic, Inc., Burlington, North Carolina
  - Neem Research Group of Charlotte, Charlotte, North Carolina
  - Bland Clinic, PA, Greensboro, North Carolina
  - Triad Clinical Trials, LLC, Greensboro, North Carolina
  - Private Practice, Raleigh, North Carolina
  - Crescent Medical Research, Salisbury, North Carolina
  - Jones Family Practice, PA, Shelby, North Carolina
  - The Lipid Center, Statesville, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Frederick C. Smith Clinic R & R Research, Marion, Ohio
  - Pharmacotherapy Research Associates, INC, Zanesville, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Lion Research, Norman, Oklahoma
  - Integris Physicians Services Clinical Research, Oklahoma City, Oklahoma
  - Memorial Clinical Research, Oklahoma City, Oklahoma
  - Blair Medical Associates Inc, Altoona, Pennsylvania
  - Tri-State Medical Group, Beaver, Pennsylvania
  - Fleetwood Medical Associates, Fleetwood, Pennsylvania
  - Family Medical Associates, Levittown, Pennsylvania
  - New England Center for Clinical Research, Cranston, Rhode Island
  - Hartwell Research Group, LLC, Anderson, South Carolina
  - Low Country Internal Medicine, Charleston, South Carolina
  - Pharmacorp Clinical Trials, INC, Charleston, South Carolina
  - The Family Healthcare Center, Clinton, South Carolina
  - Columbia Clinical Research, Columbia, South Carolina
  - Med Plus South - Strand Family Practice, Garden City, South Carolina
  - DeGarmo Institute of Medical Research, Greer, South Carolina
  - Dorchester Medical Associates, Summerville, South Carolina
  - Southeastern Research Associates, Inc., Taylors, South Carolina
  - Community Research Partners, Inc., Varnville, South Carolina
  - AM Diabetes and Endocrinology Center, Bartlett, Tennessee
  - Tri-Cities Medical Research, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - ACRC Trials, Addison, Texas
  - Discover Research Inc., Beaumont, Texas
  - MW Clinical Research, Beaumont, Texas
  - Discover Research, Bryan, Texas
  - Z&Z Medical Associates/Internal Medicine Clinical Research, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - HCA Research, Houston, Texas
  - Texas Center for Drug Development, P.A., Houston, Texas
  - Leading Edge Research, PA, Irving, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - South Texas Institutes of Health, McAllen, Texas
  - Hill Country Medical Associates, New Braunfels, Texas
  - North Hills Family Practice, North Richland Hills, Texas
  - Naidu Clinic, Odessa, Texas
  - Med-Olam Clinical Research, Pasadena, Texas
  - Southwest Clinical Research Centers, LLC, Pearland, Texas
  - Diabetes & Glandular Disease Clinic , PA, San Antonio, Texas
  - Progressive Clinical Research, Bountiful, Utah
  - Utah Clinical Trials, Salt Lake City, Utah
  - Diabetes Research Center, South Burlington, Vermont
  - Northport VA Medical Center, Northport, Virginia
  - Holston Medical Group, Weber City, Virginia
  - Madrona Medical Group - Clinical Research Dept., Bellingham, Washington
  - Summit Reserach Network, LLC, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington
- Canada (6):
  - G.A. Research Associates Moncton, New Brunswick E1G 1 A7, Moncton, New Brunswick
  - T.C. Health Center, Carbonear, Newfoundland and Labrador
  - LMC Endocrinology Centres (Barrie) Ltd., Barrie, Ontario
  - LMC Endocrinology Centres -(Etobicoke) Ltd. ,, Etobicoke, Ontario
  - LMC Endocrinology Centres -(Thornhill), Thornhill, Ontario
  - LMC Endocrinology Centres (Toronto) Ltd., Toronto, Ontario
- India (6):
  - Madras Diabetes Research Foundation, Gopālapuram, Chennai
  - Medicity Hospital, Hyderabaad, Hyderabad
  - Manipal Hospital, Bangalore
  - MV Hospital for Diabetes and Diabetes Research Centre, Chennai
  - Diabetes Thyroid Hormone Research Institute Pvt Ltd., Indore
  - Christian Medical College, Vellore
- Malaysia (3):
  - University Malaya Medical Centre, Selangor Darul Ehsan, Ehsan
  - Hospital University Kebangsaan Malaysia, Kuala Lumpur, Selangor
  - Hospital Putrajaya, Selangor Darul Ehsan, Selangor
- Philippines (3):
  - Jose R. Reyes Memorial Medical Center, Sta Cruz, Manila
  - Metropolitan Medical Center, Manila
  - Institute for Studies on Diabetes Foundation, Marikina City
- Puerto Rico (5):
  - Policlinica Dr. Luis Rodriguez Carrasquillo, Carolina
  - Yolanda Sierra Medical Office, Levittown
  - Endocrine Lipid Diabetes Research Institute, Ponce
  - Centro Clinico San Patricio, San Juan
  - Miguel Sosa-Padilla, M.D., San Juan
- Romania (5):
  - CMI Cardiologie, Baia Mare
  - Paulescu Institute, Bucharest
  - Anamed SRL, Oradea
  - Emergency County Hospital Ploiesti, Ploieşti
  - Policlinica, Timișoara
- Slovakia (7):
  - Diabetologicka ambulancia, Komarnanska, Velky Meder
  - Zeleznicne zdravotnictvo s.r.o., Diabetologicka ambulancia, Košice
  - Diabetologicka ambulancia, Nové Mesto nad Váhom
  - Diabetologicka ambulancia, Prešov
  - Mestska poliklinika Sered, Diabetologicka ambulancia, Sereď
  - Diabetologicka ambulancia, Šahy
  - Diabetologicka ambulancia, Trebišov

REFERENCES:
- See also: Results for CLAF237B2201 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4586